CLINICAL TRIAL: NCT02633878
Title: Chinese Herbal Medicine (New "Shoutai Wan") and/or Oral Progesterone Intervention Trial for Threatened Miscarriage (CHOP-IT): An International Cooperative Multicenter Randomized Controlled Trial
Brief Title: Chinese Herbal Medicine (New "Shoutai Wan") and/or Oral Progesterone Intervention Trial for Threatened Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Director of Obstetrics and Gynecology Department, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHOP-IT
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Threatened Miscarriage
Keywords: Threatened Miscarriage; Micronized Progesterone; Chinese Herbal Medicine; Live Birth
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NSTW + OP (Experimental): NSTW one pack twice daily until 12 weeks of gestations (max 84 days); OP 100 mg thrice daily until 12 weeks of gestations (max 84 days).
  Interventions: Drug: Chinese Herbal Medicine (New "Shoutai Wan") plus Oral Progesterone
- NSTW + OP placebo (Experimental): NSTW one pack twice daily until 12 weeks of gestations (max 84 days); OP Placebo 100 mg thrice daily until 12 weeks of gestations (max 84 days).
  Interventions: Drug: Chinese Herbal Medicine (New "Shoutai Wan") plus Oral Progesterone Placebo
- NSTW Placebo + OP (Experimental): NSTW Placebo one pack twice daily until 12 weeks of gestations (max 84 days); OP 100 mg thrice daily until 12 weeks of gestations (max 84 days).
  Interventions: Drug: Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo) plus Oral Progesterone
- NSTW Placebo + OP Placebo (Placebo Comparator): NSTW Placebo one pack twice daily until 12 weeks of gestations (max 84 days); OP Placebo 100 mg thrice daily until 12 weeks of gestations (max 84 days).
  Interventions: Drug: Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo) plus Oral Progesterone Placebo

INTERVENTIONS:
Drug: Chinese Herbal Medicine (New "Shoutai Wan") plus Oral Progesterone — Chinese Herbal Medicine (New "Shoutai Wan", one pack twice daily) + Oral Progesterone (100 mg thrice daily)
  Arms: NSTW + OP
Drug: Chinese Herbal Medicine (New "Shoutai Wan") plus Oral Progesterone Placebo — Chinese Herbal Medicine (New "Shoutai Wan", one pack twice daily) + Oral Progesterone Placebo (100 mg thrice daily)
  Arms: NSTW + OP placebo
Drug: Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo) plus Oral Progesterone — Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo, one pack twice daily) + Oral Progesterone (100 mg thrice daily)
  Arms: NSTW Placebo + OP
Drug: Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo) plus Oral Progesterone Placebo — Chinese Herbal Medicine Placebo (New "Shoutai Wan" placebo, one pack twice daily) + Oral Progesterone Placebo (100 mg thrice daily)
  Arms: NSTW Placebo + OP Placebo

SUMMARY:
Threatened miscarriage is manifested by vaginal bleeding, with or without abdominal pain, while the cervix is closed and the fetus is viable and inside the uterine cavity. Threatened miscarriage is a common complication of pregnancy occurring in 20% of all clinically recognized pregnancies and about half of these will eventually result in pregnancy loss. The goal of this two by two factorial, placebo controlled randomized trial is to determine that two oral medications and their combination, will mostly likely result in live birth in women with threatened miscarriage. We will evaluate the efficacy and safety of Chinese herbal medicine (New "Shoutai Wan", NSTW) and/or oral micronized progesterone (OP) for treating threatened miscarriage in this trial. Our primary outcome of this trial is live birth. We hypothesize that: 1. treatment with NSTW plus OP or OP placebo is more likely to result in live birth than NSTW placebo plus OP or placebo; 2. treatment with OP plus NSTW or NSTW placebo is more likely to result in live birth than OP placebo plus NSTW or NSTW placebo; 3. treatment with combination of NSTW and OP is more likely to result in live birth than combination of NSTW placebo and OP placebo.

DETAILED DESCRIPTION:
The causes of spontaneous miscarriage are diverse and comprise chromosomal, genetic, anatomical, immunological, hormonal, infectious and psychological factors, the other factors contribute to an increased risk include advancing paternal and maternal age and mothers with systemic diseases, such as diabetes or thyroid dysfunction. The incidence is difficult to determine precisely because it occurs very early during a pregnancy and almost 30% of early pregnancy may go unrecognized; the pathogenesis of pregnancy loss in this condition is still remains obscure. Compared with healthy women, the women with threatened miscarriage were found not only to have increased rate of antepartum haemorrhage, prelabour rupture of the membranes, preterm delivery, and intrauterine growth restriction, but also suffer from significant psychological impairment including considerable anxiety and stress, depression, sleep disturbances, anger, and marital disturbances.

To date, therapies have limited effectiveness in treating threatened miscarriage and are empirical. Bed rest does not prevent pregnancy loss. Acetaminophen may have some effects on relieving pain only. The most commonly used prescription medication was human chorionic gonadotropin (hCG), maintaining the luteotrophic effects to support continued secretion of estrogen and progesterone, but it's beneficial effects still cannot be verified. Progesterone is another most commonly used standard medication, maintaining the endometrial proliferation and preventing poor decidualization. A number of recent studies in women with threatened miscarriage shown a reduction in pregnancy loss with progesterone treatment. But progestogens are a group of hormones, including both the natural female sex hormone progesterone and the synthetic forms. Micronized progesterone is a kind of progesterone; it is structurally and pharmacologically very similar to natural progesterone and has good oral bioavailability. It is especially suitable for women with threatened miscarriage as it does not have androgenic or oestrogenic effects on the foetus. A recent review of maternal use of micronized progesterone during pregnancy also found no evidence for an increased risk of congenital malformations. However it may only be suitable to treat women with threatened miscarriage who have low progesterone levels due to corpus luteum deficiency at the first trimester of pregnancy. There is no evidence to show the beneficial effects of progesterone to treat threatened miscarriage due to others factors. At the same time, progesterone treatment is also expensive. New or adjuvant treatments that are suitable, readily accessible, affordable, and safe are needed to treat women with threatened miscarriage.

ELIGIBILITY:
Inclusion criteria:

1. Age of women between 20-37 years.
2. Pregnant. The fetus is viable inside the uterine cavity during early pregnancy (5-10 week gestations) by ultrasound and/or serum hCG changes.
3. Bleeding symptoms: vaginal bleeding with or without abdominal pain, while the cervix is closed in during speculum examination.

Exclusion criteria:

1. Multiple pregnancies (more than one gestational sac or fetal pole in ultrasonography).
2. Ectopic pregnancy. We will define an ectopic pregnancy as any suspected adnexal mass or large amounts of free fluid in the pelvis without an accompanying intrauterine pregnancy.
3. Pregnancies of Unknown Location (PUL). This will include pregnancies with an hCG level >2500mIU/mL without visualization of an intrauterine or extrauterine (i.e. ectopic) pregnancies.
4. Non-viable pregnancy. We will define a non-viable pregnancy as: (1) an intrauterine pregnancy with a fetal pole without visualized fetal heart motion (>49 days); (2) a gestational sac>20 mm in any diameter without a yolk sac; (3) absence of a normal gestational sac at 5 weeks of pregnancy, absence of a yolk sac at 5.5-6 weeks of pregnancy, or absence of cardiac activity at 7 weeks of pregnancy by ultrasound; (4) falling serum hCG values on serial visits or between baseline and randomization visit, or serial serum hCG levels which show a plateau (2-day increase ≤ 10%).
5. Intrauterine abnormalities or submucosal fibroids distorting uterine cavity (as assessed by ultrasound).
6. Bleeding attributed to a vulvar, vaginal, or cervical source unrelated to the pregnancy.
7. For this threatened miscarriage, use of the same or similar Chinese medicine and/or progesterone more than one week.
8. History of a congenital or acquired bleeding diathesis, i.e. Hemophilia, Von Willebrands's Disease, use of anti-coagulants, etc.
9. Presence of contributing major medical disorders (regardless of severity). These include poorly controlled diabetes, uncontrolled hypertension, systemic lupus erythematosus (SLE), untreated or active cancer (any cancer in remission or non-melanoma skin cancer is not included in the exclusion criteria), liver disease, renal disease, rheumatoid arthritis, cardiac disease, pulmonary disease other than mild asthma, neurologic disease requiring medical treatment, uncontrolled hypothyroidism, uncontrolled seizure disorder. Untreated vitamin B12 deficiency, severe anemia (hct < 30%), hemophilia, gout, nasal polyps.
10. Known current or recent alcohol abuse or illicit drug use.
11. Known abnormal parental karyotype.
12. Unwilling to give informed consent.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1656 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth | At or beyond 20 completed weeks' gestation
  Rate of live birth at or beyond 20 completed weeks' gestation

SECONDARY OUTCOMES:
Pregnancy outcome: Ongoing pregnancy | Beyond 12 weeks' gestation
  Rate of ongoing pregnancy (beyond 12 weeks' gestation)
Pregnancy outcome: Miscarriage during the first trimester | During the first trimester (at or before 12 weeks' gestation)
  Rate of miscarriage during the first trimester (at or before 12 weeks' gestation)
Pregnancy outcome: Miscarriage during second and third trimesters | During second and third trimesters (beyond 12 weeks' gestation until 20 weeks)
  Rate of miscarriage during second and third trimesters (beyond 12 weeks' gestation until 20 weeks)
Pregnancy outcome: Termination | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of termination at any time during treatment and follow-up period
Pregnancy outcome: Stillbirth | At or beyond 20 weeks' gestation
  Rate of stillbirth (at or beyond 20 weeks' gestation)
Pregnancy outcome: Induced abortion | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of induced abortion at any time during treatment and follow-up for any reasons
Pregnancy outcome: Gestational age at delivery | Up to 1 day after delivery
  Gestational age at delivery (weeks and days)
Pregnancy outcome: Preterm birth | Birth before 37 completed weeks' gestation (up to and including 36 weeks and 6 days of gestation)
  Rate of preterm birth (birth beyond 28 week and before 37 completed weeks' gestation (up to and including 36 weeks and 6 days of gestation))
Pregnancy outcome: Extreme preterm birth | Birth beyond 20 weeks and before 28 completed weeks' gestation (up to and including 27 weeks and 6 days of gestation)
  Rate of extreme preterm birth (birth beyond 20 weeks and before 28 completed weeks' gestation (up to and including 27 weeks and 6 days of gestation))
Pregnancy outcome: Full-term birth | At or beyond 37 weeks' gestation, and before 42 weeks' gestation
  Rate of full-term birth (at or beyond 37 weeks' gestation, and before 42 weeks' gestation)
Pregnancy outcome: Post-term birth | At or beyond 42 weeks' gestation
  Rate of post-term birth (at or beyond 42 weeks' gestation)
Neonatal outcome: Birth weight | When neonatal is born
  Birth weight of neonatal (adjusted for gestational age and sex by Chinese standards)
Neonatal outcome: Small for gestational age | When neonatal is born
  Rate of small for gestational age when neonatal is born
Neonatal outcome: Large for gestational age | When neonatal is born
  Rate of large for gestational age when neonatal is born
Neonatal outcome: Congenital malformation | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of congenital malformation
Other outcome: Mean score change in TCM Symptom Questionnaire | From date of randomization until the date of end of treatment, assessed up to 2 months
  Mean score change in TCM Symptom Questionnaire from baseline to the end of intervention. The questionnaire covers many dimensions including symptoms (amount of vaginal bleeding, severity of abdominal pain and other general symptoms), emotional factors and so on. The minimum and maximum value are depend on the symptoms of the patient respectively.
Other outcome: Mean score change in 12-Item Short-Form Health Survey | From date of randomization until the date of end of treatment, assessed up to 2 months
  Mean score change in 12-Item Short-Form Health Survey from baseline to the end of intervention. The minimum value is 0 and the maximum value is 100, and higher scores mean a better outcome.
Other outcome: Mean score change in Self-Rating Anxiety Scale | From date of randomization until the date of end of treatment, assessed up to 2 months
  Mean score change in Self-Rating Anxiety Scale from baseline to the end of intervention. The minimum value is 20 and the maximum value is 80, and lower scores mean a better outcome.

OTHER OUTCOMES:
Safety outcomes: Serious adverse events - Acute kidney injury (AKI) | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of acute kidney injury (AKI)
Safety outcomes: Serious adverse events - Drug induced liver injury (DILI) | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of drug induced liver injury (DILI)
Safety outcomes: Serious adverse events - Hospitalization | At any time during treatment (up to 2 months) and follow-up period (up to 1 year)
  Rate of hospitalization (for threatened abortion in second and third trimester of pregnancy, hyperemesis gravidarum, aggravation-vaginal bleeding, cervical polypectomy, fall injuries and other reasons)
Safety outcomes: Adverse events - Nausea and vomiting | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of nausea and vomiting.
Safety outcomes: Adverse events - Dizziness | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Dizziness.
Safety outcomes: Aadverse events - Fetal and neonatal complications | From date of randomization until the date of end of pregnancy
  Rate of fetal and neonatal complications. Fetal complications including distress, and neonatal complications including early infection, NICU admission, pneumonia, hyperbilirubinemia.
Safety outcomes: Adverse events - Fatigue | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Fatigue.
Safety outcomes: Adverse events - Anorexia | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Anorexia.
Safety outcomes: Adverse events - Constipation | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Constipation.
Safety outcomes: Adverse events - Breast distention and pain | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Breast distention and pain
Safety outcomes: Adverse events - Upper respiratory tract infection | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Upper respiratory tract infection.
Safety outcomes: Adverse events - Abdominal pain | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Abdominal pain
Safety outcomes: Adverse events - Somnolence | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Somnolence
Safety outcomes: Adverse events - Insomnia | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Insomnia
Safety outcomes: Adverse events - Anemia | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Anemia
Safety outcomes: Adverse events - Diarrhea | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Diarrhea
Safety outcomes: Adverse events - Suspected acute kidney injury (AKI) | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Suspected acute kidney injury (AKI)
Safety outcomes: Adverse events - Suspected drug-induced liver injury (DILI). | From date of randomization until the date of end of treatment, assessed up to 2 months.
  Rate of Suspected drug-induced liver injury (DILI).
Safety outcomes: Maternal complications - Pregnancy induced hypertension | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Pregnancy induced hypertension
Safety outcomes: Maternal complications - Pre-eclampsia | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Pre-eclampsia
Safety outcomes: Maternal complications - Gestational diabetes mellitus | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Gestational diabetes mellitus
Safety outcomes: Maternal complications - Placenta previa | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Placenta previa
Safety outcomes: Maternal complications - Pre-labour rupture of membranes | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Pre-labour rupture of membranes
Safety outcomes: Maternal complications - Postpartum haemorrhage | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Postpartum haemorrhage
Safety outcomes: Fetal complications - Fatal distress | From the date of end of treatment until the date of end of pregnancy, assessed up to 34 weeks.
  Rate of Fatal distress
Safety outcomes: Neonatal complications - Neonatal Early infection | From the date of delivery, assessed up to 6 weeks
  Rate of Neonatal Early infection
Safety outcomes: Neonatal complications - Neonatal NICU admission | From the date of delivery, assessed up to 6 weeks
  Rate of Neonatal NICU admission
Safety outcomes: Neonatal complications - Neonatal pneumonia | From the date of delivery, assessed up to 6 weeks
  Rate of Neonatal pneumonia
Safety outcomes: Neonatal complications - Neonatal hyperbilirubinemia | From the date of delivery, assessed up to 6 weeks
  Rate of Neonatal hyperbilirubinemia

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ke Wu, Ph.D, Study Chair — First Affiliated Hospital of Heilongjiang Chinese Medicine University
Locations (22):
- China (22):
  - The First Affiliated Hospital of Anhui University of Chinese Medicine, Hefei, Anhui
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Da Qing Long Nan Hospital, Daqing, Heilongjiang
  - First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Luoyang Hospital of Traditional Chinese Medicine, Luoyang, Henan
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Changzhou Hospital of Traditional Chinese Medicine, Changzhou, Jiangsu
  - Suqian Maternity Hospital, Suqian, Jiangsu
  - The People's Hospital of Siyang, Suqian, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xuzhou Maternal and Child Health Hospital, Xuzhou, Jiangsu
  - Jiangxi Maternity and Child Health Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi
  - Dalian Maternal and Child Health Hospital, Dalian, Liaoning
  - Dalian women and children's medical group, Dalian, Liaoning
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Ningxia Chinese Medicine Research Center, Yinchuan, Ningxia
  - Taian City Central Hospital, Tai’an, Shandong
  - Shanxi Traditional Chinese Medical Hospital, Taiyuan, Shanxi
  - Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Wenzhou TCM Hospital of Zhejiang Chinese Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No